CLINICAL TRIAL: NCT06897228
Title: A Single-center, Single-arm, Dose-escalation Exploratory Clinical Trial on the Safety and Efficacy of PANK-003 Cell Injection Combined with Standard Adjuvant Chemotherapy After Surgery in Patients with Solid Tumors
Brief Title: PANK-003 Cell Injection Combined with Standard Adjuvant Chemotherapy After Surgery in Patients with Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Celconta Life Science Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024YP01H01
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumors, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PANK-003 cell injection combined with standard postoperative adjuvant chemotherapy (Experimental): PANK-003 cell injection combined with standard postoperative adjuvant chemotherapy
  Interventions: Drug: PANK-003 cell injection

INTERVENTIONS:
Drug: PANK-003 cell injection — PANK-003 cell injection

SUMMARY:
A single-center, single-arm, dose-escalation exploratory clinical trial on the safety and efficacy of PANK-003 cell injection(Peripheral blood-derived allogeneic natural killer cells )combined with standard adjuvant chemotherapy after surgery in patients with solid tumors

DETAILED DESCRIPTION:
This project is a prospective, single-arm, open-label, single-dose, multiple-administration dose-finding study, which aims to evaluate the safety, tolerability, and efficacy characteristics of the PANK-003 cell preparation in subjects after adjuvant chemotherapy following surgery for solid tumors.

The study will enroll subjects with pathologically diagnosed solid tumors (lung cancer, esophageal cancer, gastric cancer, breast cancer) who have received adjuvant chemotherapy after surgical treatment or after neoadjuvant therapy plus surgical treatment.

The study includes a screening period, a treatment period, and an observation and follow-up period.

The main objectives :

To evaluate the safety and tolerability of multiple injections of PANK-003 cell injection combined with standard postoperative adjuvant chemotherapy in the treatment of patients with solid tumors.

The secondary objectives :

To preliminarily evaluate the efficacy of multiple injections of PANK-003 cell injection combined with standard postoperative adjuvant chemotherapy in the treatment of patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign the informed consent form;
2. At the time of screening, the age should be between 18 and 75 years old (inclusive), regardless of gender;
3. Patients who have been histologically confirmed or diagnosed by imaging (computed tomography (CT) examination, magnetic resonance imaging (MRI) examination or positron emission tomography (PET) scan CT (PET/CT)) as postoperative patients with malignant solid tumors;
4. Patients who have undergone surgical treatment and are going to receive or are currently undergoing postoperative adjuvant chemotherapy;
5. At the time of enrollment, the expected survival time is more than 6 months;
6. The Eastern Cooperative Oncology Group (ECOG) performance status score is 0 or 1;
7. At the time of screening, the laboratory tests should meet the following requirements:

   * White blood cell count ≥ 3.0×10⁹/L;
   * Neutrophil count ≥ 1.5×10⁹/L;
   * Lymphocyte count ≥ 0.5×10⁹/L;
   * Hemoglobin ≥ 90 g/L;
   * Platelets ≥ 75×10⁹/L;
   * Serum total bilirubin ≤ 2.0× the upper limit of normal value (ULN). For patients with a history of Gilbert's syndrome/suspected of having the disease, the total bilirubin (TBIL) should be ≤ 3×ULN;
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5× ULN;
   * Creatinine < 1.5×ULN and endogenous creatinine clearance rate ≥ 50 mL/minute (Cockcroft-Gault method for calculating creatinine clearance rate: For men, creatinine clearance rate = [(140 - age) × body weight (kg)] / [0.818 × creatinine (μmol/L)]; For women, creatinine clearance rate = [(140 - age) × body weight (kg) × 0.85] / [0.818 × creatinine (μmol/L)]);
8. Good lung function, with a baseline fingertip pulse oximetry saturation ≥ 95% in an indoor air environment;
9. Female subjects of childbearing age must undergo a serum pregnancy test at the time of screening with a negative result, and be willing to use a medically approved highly effective contraceptive method during the study period and for at least 1 year after the last study treatment. For male subjects whose partners are of childbearing age, they should have undergone surgical sterilization or agree to use an effective contraceptive method during the study period and for at least 1 year after the last study treatment;
10. Be evaluated by the investigator as suitable for inclusion in this clinical study.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Individuals with a history of allergy to any component of the cell product;
3. Patients with other malignant tumors, except for the following situations: cured non-melanoma skin cancer, in-situ cervical cancer, localized prostate cancer, superficial bladder cancer, and other malignant tumors with a disease-free survival period of more than 5 years;
4. Positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg), positive for hepatitis B e antibody (HBe-Ab) and/or hepatitis B core antibody (HBc-Ab), and the HBV-DNA copy number is greater than the lower limit of measurability; positive for hepatitis C antibody (HCV-Ab); positive for Treponema pallidum antibody (TP-Ab); positive for human immunodeficiency virus (HIV) antibody test; anyone meeting any one of these items;
5. Patients who have received drugs from other clinical trials or other cellular immunotherapies within 28 days before the screening period;
6. Those who have received live vaccines or live attenuated vaccines within 4 weeks before NK cell infusion;
7. Patients with comorbidities that, in the judgment of the investigator, require treatment with systemic corticosteroids or other immunosuppressive drugs during the study period;
8. Individuals with a high allergic constitution, those allergic to any component of the NK preparation product, including those allergic to serum albumin; those allergic to commonly used emergency and anesthetic drugs;
9. Having any unstable circulatory system diseases within 180 days before screening, including but not limited to unstable angina pectoris, myocardial infarction, heart failure [New York Heart Association (NYHA) class ≥ III], severe arrhythmia requiring drug treatment, or having undergone angioplasty, coronary artery stent implantation, or coronary artery bypass grafting within 180 days before screening;
10. Diseases or other situations that the investigator deems unsuitable for this clinical study (such as high allergic constitution, poorly controlled diabetes mellitus, uncontrolled infections, presence of central nervous system diseases, bleeding and thrombotic tendencies; as well as poor compliance, drug abuse, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 21 days after the completion of a single administration
  Dose limiting toxicity (DLT) in the dose escalation phase
Incidence of Treatment Related adverse events (AEs) | 1 year
  Incidence of Treatment Related AEs, AEs of special interest
Maximum tolerated dose (MTD) | 21 days after the completion of a single administration
  Maximum tolerated dose (MTD) in the dose escalation phase

SECONDARY OUTCOMES:
Evaluate the disease - free survival (DFS) | 1 year
  The time from the date of first administration of PANK-003 cell injection to tumor recurrence or death from any cause
Evaluate the overall survival (OS) | 1 year
  The time from the date of first administration of PANK-003 cell injection to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- AnYang Tumor Hospital, Anyang, Henan, China

IPD SHARING:
Plan to Share IPD: No